CLINICAL TRIAL: NCT04562454
Title: An Exploratory Study on the Application of Continuous Glucose Monitoring System in the Measurement of Individual Glycemic Index After Eating Different Diets
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20200920-JS-2450
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal group (Experimental): Specific diet with CGM for 5days
  Interventions: Other: Specific diet
- T1DM group (Experimental): Specific diet with CGM for 5days
  Interventions: Other: Specific diet
- T2DM group (Experimental): Specific diet with CGM for 5days
  Interventions: Other: Specific diet
- other type of diabetes group (Experimental): Specific diet with CGM for 5days
  Interventions: Other: Specific diet

INTERVENTIONS:
Other: Specific diet — use a specific diet in different days with CGM to konw GI of different food in diabetes

SUMMARY:
The glycemic index (GI) is used to evaluate the level of elevated blood sugar immediately after carbohydrate intake and is a classified indicator of the glycemic potential of carbohydrate-containing test foods relative to reference foods. At present, more and more clinical studies have proved that a low-GI diet is beneficial to health, and can improve blood glucose control, weight and blood lipid levels in patients with type 1 diabetes mellitus (T1DM) and type 2 diabetes mellitus (T2DM). GI is currently widely used to provide guidance on food choices for people with diabetes. However, there are great differences in blood glucose response among different individuals after eating the same food, which is related to a variety of factors，including individual gastrointestinal digestion and absorption rate,islet function,insulin resistance and region. A large number of foreign studies suggest that race affects the determination of GI, but different regions of our country have different dietary culture and different ability to digest and absorb different foods. Therefore, the traditional GI reference value does not necessarily fully reflect the blood glucose response of diabetic patients after eating a food. In this study, continuous blood glucose monitoring was carried out through CGM to monitor the overall fluctuation level of blood glucose, the time to peak and the range of blood glucose fluctuation after eating specific foods, and to obtain individual GI, after eating different diets to guide the future diet.

DETAILED DESCRIPTION:
In this study, subjects with diabetes or impaired glucose tolerance were given continuous glucose monitoring (CGM) for 3 consecutive days, given a standard meal containing 50g carbohydrates and foods to be tested for GI. The purpose of this study was to explore the fluctuation of blood glucose, the time and range of blood glucose peak after eating different diets, and to guide the individual dietary choices of the subjects. And try to find the best time and dose of hypoglycemic strategy for subjects during meals. At the same time, during the follow-up period, we observed whether the subjects could achieve better blood glucose control after adjusting their diet according to the GI of different foods. At the same time, the GI results of the same food were compared between people with normal glucose metabolism and those with abnormal glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. the experimental group: patients with diabetes or impaired glucose tolerance diagnosed clinically according to the World Health Organization's (WHO) diagnostic criteria of diabetes in 1999; the control group: according to the participants of the experimental group, matched the people with normal glucose metabolism in sex, age and region.
2. Age: 18-80 years old; 3) patients or family members who can understand the research plan and are willing to participate in this study and sign a written informed consent form and questionnaire

Exclusion Criteria:

1. severe acute complications of diabetes (diabetic ketoacidosis, hyperglycemia and hyperosmotic state, diabetic lactic acidosis) in the past 6 months;
2. serious chronic complications of diabetes, such as peripheral vascular disease leading to amputation or chronic foot ulcers, end-stage renal disease, etc., the researchers do not think it is suitable to participate in this study.；
3. patients with two or more episodes of severe hypoglycemia in the past year (such as disturbance of consciousness caused by hypoglycemia, coma, etc.), or severe unconscious hypoglycemia;
4. patients with severe impairment or circulatory disturbance of cardiac function (NYHA grade III or above), liver function (ALT, AST or TBil above the upper limit of the normal value), renal function (serum creatinine above the upper limit of the normal value) or circulatory disturbance.；
5. patients with mental illness, confusion and inability to take care of themselves;
6. patients with gastrointestinal diseases;
7. patients or their families cannot understand the conditions and objectives of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
fluctuation of blood glucose after eating different food | baseline
  use the CGM to get the area under the curve of blood glucose of different food

CONTACTS AND LOCATIONS:
Overall Officials: Weigang Zhao, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No